CLINICAL TRIAL: NCT03057119
Title: Feasibility of Screening, Brief Intervention, Referral to Treatment With Peer Navigation (SBIRT-PN) for Underserved HIV+ Adults 50+ in Primary Care Settings.
Brief Title: Feasibility of SBIRT-PN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nicole Ennis, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB201701252 - N; 1K23DA039769-01 (NIH); KL2TR001429 (NIH); OCR25582 (Other: UF OnCore)
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Substance Use; HIV/AIDS; Older Adults; Behavioral Intervention; Infectious Disease
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: A repeated measures randomized control trial design to compare patient outcomes at baseline as well as 3 and 6 months post-intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIRT Intervention (Experimental): The interventionist will discuss substance use and misuse, HIV, and the interaction of aging and substance use; will give the patient feedback on their NM-ASSIST score and assess the patient's readiness to change based on Prochaska's stages of change; motivational interviewing techniques to identify the patients' most salient reasons for addressing substance use issues. Identifying and prioritizing need; problem-solving techniques to help patients identify which services may best help them work towards their goals; will use a referral resource guide to provide the contact information of agency representatives and help the patient formulate a plan for follow-up.
  Interventions: Behavioral: Psycho-educational content (5 Minutes); Behavioral: Readiness Assessment (10 minutes); Behavioral: Goal-Setting (5 minutes); Behavioral: Identifying and prioritizing needs (5 minutes); Behavioral: Explanation of Peer Navigator and Session wrap (5 minutes)
- Treatment as Usual (No Intervention): Participants in the enhanced care treatment as usual group will receive the same illustrated handout depicting their substance use screening score and the same referral resource guide provided to those in the control group. These will be provided with only a quick introduction by the research assistant to minimize intervention elements in the control condition and to resemble the notification and referral strategy that would be standard care.

INTERVENTIONS:
Behavioral: Psycho-educational content (5 Minutes) — The interventionist will discuss substance use and misuse and the influence of substance use on self care.
  Arms: SBIRT Intervention
Behavioral: Readiness Assessment (10 minutes) — The interventionist will give the patient feedback on their ASSIST score and assess the patient's readiness to change based on Prochaska's stages of change.
  Other Names: Prochaska's stages of change.
  Arms: SBIRT Intervention
Behavioral: Goal-Setting (5 minutes) — The interventionist will use motivational interviewing techniques to identify the patients' most salient reasons for addressing substance use issues.
  Arms: SBIRT Intervention
Behavioral: Identifying and prioritizing needs (5 minutes) — The interventionist will use problem-solving techniques to help patients identify which services may best help them work towards their goals. Services will include (but are not limited to) emergency crisis services, counseling to deal with substance use, referral to local self-help groups (Alcoholics Anonymous, Narcotics Anonymous, etc.), legal assistance, faith-based counseling, mental health counseling or inpatient substance use treatment.
  Arms: SBIRT Intervention
Behavioral: Explanation of Peer Navigator and Session wrap (5 minutes) — The interventionist will use a referral resource guide to provide the contact information of agency representatives and help the patient formulate a plan for follow-up.
  Arms: SBIRT Intervention

SUMMARY:
Substance misuse is a common problem among HIV+ individuals. Research suggests that a Screening, Brief Intervention, and Treatment (SBIRT) model can be effective in reducing substance misuse in the general older adult population; however these findings have not been verified in the more vulnerable HIV+ older adult population. The present study seeks to address the problem of substance misuse in older HIV+ adults by piloting a SBIRT model for older HIV+ adults in a in a primary care setting. Individual reductions in alcohol and drug use can have significant effects on public health and safety when observed over a large population at risk for substance use problems. With wider dissemination statewide, a relatively low-cost intervention such as SBIRT could offer demonstrated benefits in this population.

DETAILED DESCRIPTION:
The current project will pilot SBIRT with a peer navigator (SBIRT-PN) versus treatment at usual (TAU) to increase substance use treatment engagement among HIV-positive adults aged 50 years and older. The investigators will recruit patients from the Southern HIV and Alcohol Research Consortium (SHARC) HIV primary care clinic network.

In order to develop effective substance use intervention models for HIV care settings the specific aims of the current project are:

Aim1: Examine the feasibility of the SBIRT-PN model at the UF Health Infectious Disease-Medical Specialties Clinic. The investigators hypothesize that the SBIRT-PN model will demonstrate high feasibility within the UF Health Infectious Disease - Medical Specialties Clinic.

Aim2a: Assess the acceptability of SBIRT-PN. The investigators hypothesize that SBIRT-PN will demonstrate high acceptability among patients enrolled in this condition.

Aim2b: Assess the acceptability of SBIRT-PN among HIV-positive individuals by age cohort (younger vs older). The investigators hypothesize that SBIRT-PN will demonstrate higher acceptability among older HIV-positive patients enrolled in this condition.

Aim3: Assess influence of SBIRT-PN model on treatment engagement and substance use compared to enhanced treatment as usual (TAU).The investigators hypothesize that those in the SBIRT-PN condition will evidence greater treatment engagement and a reduction in substance use.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care at an Infectious disease Medical Clinic
* HIV-positive (seropositive confirmed by medical records)
* have a substance misuse screening score indicating moderate or high risk.

Exclusion Criteria:

* lack fluency in English
* are unwilling to provide information for follow-up
* plan to leave the area within 6 months
* already have a referral to treatment from another provider
* unable to provide informed consent due to cognitive impairment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ennis, PHD, Principal Investigator — Florida State University
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - CAN Community Health, Jacksonville, Florida
  - Department of Health in Columbia County",, Lake City, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: SBIRT Intervention (Pre-COVID-19): Interventionist will discuss substance use/misuse, HIV, interaction of aging & substance use; give feedback on ASSIST scores; assess patients' readiness to change based on Prochaska's stages of change; motivational interviewing techniques to identify patients' most salient reasons for addressing substance use; Identify/prioritize need; problem-solving techniques to help patients identify which services may best help them work toward their goals; use referral guide to provide contact information of agency representatives & help patients formulate follow-up plan.
  Psycho-educational content: Interventionist will discuss substance use/misuse & influence of substance use on self care.
  Readiness Assessment: Interventionist will give feedback on ASSIST score & assess patients' readiness to change based on Prochaska's stages of change.
  Goal-Setting: Interventionist will use MI techniques to identify patients' most salient reasons for addressing substance use.
  Identifying/prioritizing needs: Interventionist will use problem-solving techniques to help patients identify which services may best help them work toward their goals (e.g., as crisis services, substance use counseling, local self-help groups (AA, NA, etc), legal aid, faith-based counseling, mental health counseling, or inpatient SUD treatment).
  Explanation of PN/Session wrap: Interventionist will use referral guide to provide contact information of agency representatives & help patients formulate follow-up plan.
- Phase I: Treatment as Usual (Pre-COVID-19): Participants in the enhanced care treatment as usual group will receive the same illustrated handout depicting their substance use screening score and the same referral resource guide provided to those in the control group. These will be provided with only a quick introduction by the research assistant to minimize intervention elements in the control condition and to resemble the notification and referral strategy that would be standard care.
- Phase II: CAN Pandemic Telesurvey (Post-COVID-19): Given the need for social support among people living with HIV during the COVID-19 pandemic, we made the decision to initiate a pandemic telehealth assessment that used screening, brief intervention, and referral to treatment to address behavioral and emotional distress in a among people living with at CAN Community Health, which is in the only EHE designated county in North Florida (Duval County, FL).
  Participants were asked to complete an online survey via Qualtrics at T1, T2, and T3 with the help of a research assistant affiliated with the clinic. Each survey included the Patient Health Questionnaire (PHQ-9) and Pandemic Stress Index (PSI). Participants were also asked demographic questions (e.g., about their employment), about their alcohol, tobacco, and substance use prior to and during the COVID-19 pandemic, and questions about access to (and availability of) healthcare resources.
Period: Overall Study
Arm/Group | Phase I: SBIRT Intervention (Pre-COVID-19) | Phase I: Treatment as Usual (Pre-COVID-19) | Phase II: CAN Pandemic Telesurvey (Post-COVID-19)
Started | 17 | 17 | 52
Completed T1 | 17 | 17 | 45
Completed T2 | 9 | 5 | 30
Completed T3 | 4 | 3 | 35
Completed (Completed all 3 assessments) | 4 | 3 | 13
Not Completed | 13 | 14 | 39

BASELINE CHARACTERISTICS:
Groups:
- Phase I: SBIRT Intervention (Pre-COVID-19): Interventionist will discuss substance use/misuse, HIV, the interaction of aging & substance use; give patient feedback on ASSIST score, assess patients' readiness to change based on Prochaska's stages of change; motivational interviewing techniques to identify patients' most salient reasons for addressing substance use. Identifying/prioritizing need; problem-solving techniques to help patients identify which services may best help them work toward their goals; use referral guide to provide contact information of agency representatives & help patient formulate follow-up plan
  Psychoeducational content: Interventionist will discuss substance use/misuse & the influence of substance use on self care
  Readiness Assessment: Interventionist will give patient feedback on ASSIST score & assess their readiness to change based on Prochaska's stages of change
  Goal-Setting: Interventionist will use MI techniques to identify patients' most salient reasons for addressing substance use
  Identifying/prioritizing needs: Interventionist will use problem-solving techniques to help patients identify which services may best help them work toward their goals (e.g. crisis services, counseling, local self-help groups (AA, NA, etc.), legal aid, faith-based counseling, mental health counseling or inpatient SUD tx)
  Explanation of PN/Session wrap: Interventionist will use referral guide to provide contact information of agency representatives & help the patient formulate follow-up plan
- Total: Total of all reporting groups
Arm/Group | Phase I: SBIRT Intervention (Pre-COVID-19) | Phase I: Treatment as Usual (Pre-COVID-19) | Phase II: CAN Pandemic Telesurvey (Post-COVID-19) | Total
Number analyzed (Participants) | 17 | 17 | 52 | 86
Age, Customized [Number; unit: participants]
  ≥ 50 years old | 5 | 4 | 37 | 46
  < 50 years old | 12 | 13 | 15 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 23 | 28
  Male | 15 | 14 | 29 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 15 | 16 | 0 | 31
  Unknown or Not Reported | 1 | 1 | 52 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 33 | 42
  White | 12 | 12 | 12 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Ranking Intervention as Acceptable
Description: To examine ratings of acceptability, the investigators will use the overall acceptability score and percentage of acceptability. Overall acceptability will be assessed by summing ratings from the 10-item questionnaire to provide a total intervention acceptability score for the intervention, such that acceptability scores for the intervention could range from 10 (low acceptability) to 50 (high acceptability). The intervention will be considered to have acceptability if 80% of the participants rank the intervention as acceptable (i.e., 4 or higher) on 80% or more of the scale items. The investigators will then examine each question of the Acceptability Questionnaire separately to determine strengths and weaknesses of the intervention.
Time Frame: 30 Days
Population: CAN Pandemic Telesurvey arm of this study did not include an intervention or a peer navigation element, and therefore did not have include the acceptability measures as in Phase I.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: SBIRT Intervention (Pre-COVID-19) | Phase I: Treatment as Usual (Pre-COVID-19) | Phase II: CAN Pandemic Telesurvey (Post-COVID-19)
Number analyzed (Participants) | 9 | 5 | 0
Participants | 9 | 5 |

2. Secondary Outcome: Number of Participants Who Obtained Formal Substance Use Treatment
Description: Participants will self-report if they obtained formal substance use treatment (i.e., any services sought to address substance use from individual therapy to 12 step fellowships). The investigators will request treatment facility information and permission to verify treatment. Once treatment has been verified, treatment engagement will be coded as 0= no formal treatment 1= formal treatment engagement
Time Frame: 6 Months
Population: CAN Pandemic Telesurvey arm of this study did not include an intervention or a peer navigation element, and therefore did not have include the treatment engagement measures as in Phase I.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: SBIRT Intervention (Pre-COVID-19) | Phase I: Treatment as Usual (Pre-COVID-19) | Phase II: CAN Pandemic Telesurvey (Post-COVID-19)
Number analyzed (Participants) | 17 | 17 | 0
Participants | 1 | 1 |

3. Secondary Outcome: Number of Participants Who Used Different Types of Substances (Self-Reported)
Description: A standard measure from the NIDA STTR Vulnerable Populations Data Harmonization tool kit will be used.
Time Frame: 6 Months
Population: CAN Pandemic Telesurvey arm of this study did not include an intervention or a peer navigation element, and therefore did not have include the NIDA STTR Drug and Alcohol Use Measure as in Phase I.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: SBIRT Intervention (Pre-COVID-19) | Phase I: Treatment as Usual (Pre-COVID-19) | Phase II: CAN Pandemic Telesurvey (Post-COVID-19)
Number analyzed (Participants) | 17 | 17 | 0
Participants
  Marijuana | 16 | 17 |
  Opiates/Opioids | 5 | 4 |
  Cocaine | 1 | 2 |
  Amphetamines | 0 | 1 |
  Methamphetamine | 0 | 1 |
  MDMA | 0 | 1 |

4. Secondary Outcome: Number of Participants Who Used Different Types of Substances (Biologically Confirmed Via Urinalysis)
Description: A CLIA 12-Panel Instant Drug Test Cup (CLIAwaivedTM, San Diego, CA), which tests for the presence of 12 common substances in the urine will be used.
Time Frame: 6 Months
Population: CAN Pandemic Telesurvey arm of this study did not include an intervention or a peer navigation element, and therefore did not have include the urinalysis measure as in Phase I.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: SBIRT Intervention (Pre-COVID-19) | Phase I: Treatment as Usual (Pre-COVID-19) | Phase II: CAN Pandemic Telesurvey (Post-COVID-19)
Number analyzed (Participants) | 17 | 17 | 0
Participants
  Marijuana | 16 | 17 |
  Buprenorphine | 1 | 1 |
  Methadone | 3 | 1 |
  Tricyclic Antidepressants | 4 | 7 |
  Barbiturates | 0 | 0 |
  Benzodiazepines | 4 | 2 |
  Oxycodone | 2 | 2 |
  Amphetamines | 0 | 1 |
  Methamphetamine | 0 | 1 |
  Cocaine | 1 | 2 |
  MDMA | 0 | 2 |
  PCP | 0 | 0 |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the entire study data collection process (6 months for each participant)
Arm/Group | Phase I: SBIRT Intervention (Pre-COVID-19) | Phase I: Treatment as Usual (Pre-COVID-19) | Phase II: CAN Pandemic Telesurvey (Post-COVID-19)
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/17 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/52
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/52

LIMITATIONS AND CAVEATS:
In March 2020, the COVID-19 pandemic made in-person assessments as described in Phase I (SBIRT-PN & TAU), particularly involving vulnerable populations such as PLWH and older adults, impossible. Recommendations for social distancing/self-isolation remained in place for extended periods of time. Data was needed regarding the impact of the pandemic, both physically and emotionally, on PLWH. We gathered this data within a specialized HIV care setting in order to optimize health outcomes (Phase II).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03057119/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03057119/SAP_001.pdf
  • Informed Consent Form (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT03057119/ICF_002.pdf